CLINICAL TRIAL: NCT05713760
Title: A Phase 2, Single-Arm, Open-Label, Single Center Study to Assess Efficacy and Safety of Tirbanibulin Ointment 1% in Adult Subjects With Superficial Basal Cell Carcinoma (sBCC) on the Neck, Trunk, or Extremities (Excluding Axilla, Anogenital, and Face/Scalp)
Brief Title: Proof of Concept Study to Access Superficial Basal Cell Carcinoma in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Institute for Clinical Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AICR-BCC-01
Record Dates: First submitted 2023-01-16; First posted 2023-02-06 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Superficial Basal Cell Carcinoma
MeSH Terms: interventions — tirbanibulin

STUDY DESIGN:
Intervention Model Description: Open Label Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5 Day treatment course 1 with Tirbanibulin Ointment 1% (Experimental): 10 Subjects will be given one study kit containing single-dose packets of Tirbanibulin Ointment 1% and instructed to topically apply to the treatment area once daily for 5 consecutive days.
  Interventions: Drug: Tirbanibulin Ointment 1%
- 5 Day treatment course 2 with Tirbanibulin Ointment 1% (Experimental): Subjects with unresolved lesion will be given an additional study kit containing single-dose packets of Tirbanibulin Ointment 1% and instructed to topically apply to the treatment area once daily for 5 consecutive days.
  Interventions: Drug: Tirbanibulin Ointment 1%

INTERVENTIONS:
Drug: Tirbanibulin Ointment 1% — Klisyri® ointment is a microtubule inhibitor for topical use and is currently on the market for the treatment of actinic keratosis of the face or scalp. The chemical name of tirbanibulin is N-benzyl-2-(5-(4-(2- morpholinoethoxy)phenyl)pyridin-2-yl) acetamide. Tirbanibulin ointment 1% contains 10 mg tirbanibulin per gram of white to off-white ointment containing mono- and di-glycerides and propylene glycol and is supplied in packets containing 250 mg of tirbanibulin ointment 1%. Each packet includes single-dose packets (2.5 mg tirbanibulin in 250 mg) to be applied to evenly cover up to 25 cm² of the treatment field once daily for 5 consecutive days using 1 single-dose packet per application.
  Other Names: Klisyri (tirbanibulin ointment 1%)

SUMMARY:
This is a Phase 2, Single-Arm, Open-Label, Single Center, Proof of Concept Study to Assess Efficacy and Safety of Tirbanibulin Ointment 1% in Adult Subjects with superficial basal cell carcinoma (sBCC) on the neck, trunk, or extremities (excluding, axilla, anogenital, and face/scalp).

DETAILED DESCRIPTION:
Eligible subject should have one naïve superficial basal cell carcinoma (sBCC) that will be included in the study. sBCC lesion included in the study will initially be confirmed by biopsy (either shave or punch), such that the amount of lesion remaining is at least 25% of the initial lesion surface area, and the initial lesion is at least 6mm in diameter and no more than 20mm in diameter. The total surface area of all treatment area must be <25cm squared. To minimize the burden of the subject, biopsies (either shave or punch) taken within 6 months prior to screening can be considered.

The treatment area (visible sBCC with 5mm margin of normal skin) will be marked with indelible marker (e.g., surgical marker) at Screening/Baseline (Day 1 pre-dose) at the investigational site. Lesion marking should be applied about 3~4mm from the sBCC. This will be transferred to an acetate sheet with 3 anatomical landmarks marked, Subject number, and location as well.

Approximately 10 subjects who meet the study criteria will be enrolled. The study consists of Screening, Treatment, LSR and Response Assessment and Excision Period, Suture Removal, and Follow Up. After a Screening Period of up to 29 days, subjects will return to the site for confirmation of eligibility. Eligible subjects will be randomized on Day 1 to treatment course 1 for a 5 consecutive day treatment course.

Subjects will return to the clinical site for LSR assessment, Visit 3, on day 8 and at the Response Assessment or Possible Excision, Visit 4, on day 26. If lesion is assessed as resolved, excision will be performed, Suture Removal, Visit 5, at day 36, and Follow Up, visit 6, on day 54. If lesion is assessed as not resolved at Visit 4, subjects will then proceed to Treatment Course 2 for another 5 consecutive days. For subjects who completed Treatment Course 2, subjects will return to the clinical site for LSR assessment, Visit 4a, on day 33, Response Assessment and Excision, Visit 4b, on day 51, Suture Removal, Visit 5, on day 61, and Follow Up, Visit 6, on day 79 .

The duration of the entire study from first subject, first visit to last subject, last visit is anticipated to be approximately 9 months. For the Screening, Treatment, LSR and Response Assessment and Excision Periods, Suture Removal, and Follow Up Period each subject will participate for up to 80 days:

Screen up to 29 days prior to Day 1, treatment course for 5 consecutive days with a possibility of receiving a second treatment course, LSR Assessments for 3 days, Response Assessment for 26 days, Excision, with Suture Removal 10 days from the excision, and Follow Up 28 days after excision.

Subjects will be given verbal and written instructions on self-administration and receive study drug for Treatment Course 1 including 1 study kit containing 5 daily single-dose packets, 1 for each day of treatment. The first dose will be applied by the subject under the supervision of study site personnel. Subjects will then take home the study kit containing the remaining single-dose packets of study drug for daily self-administration on the next 4 consecutive days. The written instructions will include a dosing log where the subjects will record the date and time of study drug self-administration. For subjects completing Treatment Course 2, the same instructions and dosing apply.

The Investigator may withdraw a subject from study treatment or withdraw the subject from the study at any time for safety or administrative reasons. The subject may decide to discontinue study treatment or withdraw from the study at any time for any reason. The Investigator must document the reason for discontinuing a subject from treatment or from the study if known, or why the subject withdrew consent, if applicable. Subject disposition information will be collected on the electronic case report form (eCRF).

Subjects who do not complete treatment for course 1 or 2 and withdraw from study treatment (for reasons other than death or withdrawal of consent) will be encouraged to continue the post-treatment visits. At the time of withdrawal from the study, the subject should complete the early termination assessments (Day 26 assessments).

Subjects will be instructed to contact the site to report severe or intolerable Local Skin Reactions during the treatment course(s) to schedule an Unscheduled visit for Investigator assessment of Local Skin Reactions and treatment, per Investigator judgement.

In females of childbearing potential, a urine pregnancy test will be performed at the site at the screening and baseline visit. Test results must be reviewed before randomization.

The Investigator or a qualified staff member must obtain standardized photography of the subject's treatment area at the Baseline visit, LSR and Response Assessment Periods, Excision visit, and Suture Removal visit. Additionally, photos may be captured at the Follow Up visit if the the subject has any unresolved Local Skin Reactions (LSR), and/or pigmentation and scarring in the treatment area. The photographs are to document the appearance of the subjects' treatment area and to assist with the identification and confirmation of the location of the treatment area throughout the study. Site will supply their own camera equipment for the study and photos will be uploaded to the eCRF.

Two views will be taken for each standardized photography assessment:

1. The treatment area with sBCC lesion marked with the surgical marker.
2. Close-Up of Treatment Area including a ruler with millimeter markings in the frame of the picture (not covering the lesion marked).

On the day of excision, the investigator will perform all safety and Local Skin Reaction assessments, as well as an assessment of whether the sBCC is clinically present. If the lesion is no longer clinically present, it will be assessed as a clinically complete response. After all assessments are performed, an elliptical excision will be performed per usual clinical practice on day 26 or 51 using the acetate sheet/transparency marked at screening and baseline with both the lesion margin and treatment margins (5mm beyond the lesion margin), using the 3 anatomical landmarks on the acetate/transparency to identify the lesion location. An ellipse will incorporate both the lesion and treatment margins (i.e., at least 5mm beyond the lesion margin). This specimen will be sent for pathologic review. If the pathology report fails to reveal sBCC in the excision specimen, this will be considered a pathology complete response. If the lesion achieves both clinical and pathology complete response, then it will be deemed to have achieved complete response.

All Adverse Events (AEs), regardless of relationship to study drug or procedure, should be collected beginning from the time the subject signs the study Informed Consent Form (ICF) through the final subject contact in the study. Subjects who fail screening primarily due to AE(s) must have the AE(s) recorded in the AE eCRF and screen failure reported on the eCRF. All Serious Adverse Events (SAEs) must be followed to resolution or, if resolution is unlikely, to stabilization.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old.
2. Willingness and ability to sign the informed consent form and Health Insurance Portability and Accountability Act (HIPAA) form. A study-specific informed consent form and a HIPAA form must be obtained in writing for all subjects prior to starting any study procedures.
3. Present of 1 naïve sBCC on the neck, trunk, or extremities (excluding, axilla, anogenital, and face/scalp) that:

   * is between 6 and 20mm in greatest diameter
   * >2cm from a hairline
   * Must lack any evidence of aggressive growth patterns (e.g., severe squamous metaplasia, infiltrative/desmoplastic features, or basosquamous features)
4. sBCC assessed as non-naïve (e.g., previously treated, or recurrent) or non-eligible by biopsy and at least 5cm away from an eligible lesion should be excised or treated with Electrodesiccation and Curettage (ED&C) in a timely manner.
5. Free of significant physical abnormalities (e.g., tattoos, dermatoses) within the potential treatment area plus a 5cm radius surrounding the lesion as they may interfere with examination or final evaluation, in the opinion of the investigator.
6. Willingness to stop the use of moisturizers, sunscreens, and any other cosmetics within the treatment area plus a 5cm radius from screening until final the visit.
7. Willingness to abstain from sunbathing or the use of artificial tanning from screening until the final visit. Subjects with a sunburn in the treatment area cannot be included until fully recovered.
8. Subjects must be healthy or have a medical condition that is stable in the opinion of the investigator.
9. Females must be postmenopausal (>45 years of age with at least 12 months of amenorrhea), surgically sterile (by hysterectomy, bilateral oophorectomy, or tubal ligation); or, if of childbearing potential, must be using highly effective contraception for at least 30 days or 1 menstrual cycle, whichever is longer, prior to study treatment and must agree to continue to use highly effective contraception for at least 30 days following their last dose of study treatment. Highly effective contraception includes oral hormonal contraceptives, hormonal contraceptive implant, injection or patch, intrauterine device, or complete abstinence from sexual intercourse.
10. Sexually active males who have not had a vasectomy, and whose partner is reproductively capable, must agree to use barrier contraception from Screening through 90 days after their last dose of study treatment.

Exclusion Criteria:

1. Location of the treatment area is:

   * On face, scalp, anogenital, axillae
   * Within 5 cm of an incompletely healed wound
   * Within 2 cm of hairline
2. Anticipated need for in-patient hospitalization or in-patient surgery from Day 1 to Day 57.
3. Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for Actinic Keratosis (AK) within the treatment area or within 2 cm of the treatment area, within 8 weeks prior to the Screening visit.
4. Use of the following therapies and/or medications within 2 weeks prior to the Screening visit:

   * Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the treatment area or within 2 cm of the selected treatment area
   * Acid-containing therapeutic products (e.g., salicylic acid or fruit acids, such as alpha and beta-hydroxyl acids and glycolic acids), topical retinoids, or light chemical peels within the treatment area or within 2 cm of the selected treatment area
   * Topical salves or topical steroids within the treatment area or within 2 cm of the selected treatment area
   * Artificial tanners within the treatment area or within 5 cm of the selected treatment area
5. Use of the following therapies and/or medications within 4 weeks prior to the Screening visit:

   * Treatment with immunomodulators (e.g., azathioprine), cytotoxic drugs (e.g., cyclophosphamide, vinblastine, chlorambucil, methotrexate) or interferons/interferon inducers
   * Treatment with systemic medications that suppress the immune system (e.g., cyclosporine, prednisone, methotrexate, alefacept, infliximab)
   * Use of systemic retinoids (e.g., isotretinoin, acitretin, bexarotene) within 6 months prior to the Screening visit
6. A history of sensitivity and/or allergy to any of the ingredients in the study medication.
7. A skin disease (e.g., atopic dermatitis, psoriasis, eczema) or condition (e.g., scarring, open wounds) that, in the opinion of the Investigator, might interfere with the study conduct or evaluations, or which exposes the subject to unacceptable risk by study participation.
8. Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would expose the subject to unacceptable risk by study participation.
9. Females who are pregnant or nursing.
10. Participated in an investigational drug trial during which an investigational study medication was administered within 30 days or 5 half-lives of the investigational product, whichever is longer, before dosing.
11. In the opinion of the investigator, are unable or unlikely to comply with the administration schedule and study evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Complete clearance rate of sBCC lesion | 26 days for subjects who completed 1 course of treatment and 51 days for subjects who completed 2 courses of treatment
  The primary efficacy endpoint will be the percent of subjects with both clinical and pathological clearance of sBCC lesion for subjects who completed 1 course of treatment and subjects who completed 2 courses of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research
Locations (1):
- Austin Institute for Clinical Research, Inc., Pflugerville, Texas, United States

REFERENCES:
- [Background] Blauvelt A, Kempers S, Lain E, Schlesinger T, Tyring S, Forman S, Ablon G, Martin G, Wang H, Cutler DL, Fang J, Kwan MR; Phase 3 Tirbanibulin for Actinic Keratosis Group. Phase 3 Trials of Tirbanibulin Ointment for Actinic Keratosis. N Engl J Med. 2021 Feb 11;384(6):512-520. doi: 10.1056/NEJMoa2024040. PMID 33567191
- [Result] Hong JB, Wu PY, Qin A, Huang YW, Tseng KC, Lai CY, Chan WK, Fang J, Cutler DL, Tsai TF. Topical Tirbanibulin, a Dual Src Kinase and Tubulin Polymerization Inhibitor, for the Treatment of Plaque-Type Psoriasis: Phase I Results. Pharmaceutics. 2022 Oct 11;14(10):2159. doi: 10.3390/pharmaceutics14102159. PMID 36297594